CLINICAL TRIAL: NCT00454181
Title: Evaluation of Natural Human Interferon Alpha Administered Oromucosally in the Treatment of Oral Warts in HIV-seropositive Subjects Receiving Combination Anti-retroviral Therapy: A Phase 2 Clinical Trial
Brief Title: Treatment of Oral Warts in HIV+ Patients
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Ainos, Inc. (f/k/a Amarillo Biosciences Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 03HUHI19
Record Dates: First submitted 2007-03-29; First posted 2007-03-30 (Estimated); Results first posted 2011-01-13 (Estimated); Last update posted 2011-09-16 (Estimated); Status verified 2011-09

CONDITIONS: Papillomatosis; HIV Infections
Keywords: human immunodeficiency virus; human papilloma virus; warts, oral; papillomatosis; treatment experienced
MeSH Terms: conditions — Papilloma; HIV Infections; Acquired Immunodeficiency Syndrome; Warts | interventions — Interferon-alpha; Maltose; Sugars

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- IFN lozenges (Experimental): 500 IU Interferon-alpha lozenges for oral dissolution
  Interventions: Drug: Interferon-alpha
- placebo lozenges (Placebo Comparator): 200 mg lozenges containing anhydrous crystalline maltose
  Interventions: Other: placebo

INTERVENTIONS:
Drug: Interferon-alpha — 500 IU interferon-alpha lozenges taken 3 times per day for 24 weeks
  Other Names: Veldona; IFN-alpha lozenge; low dose IFN lozenge
  Arms: IFN lozenges
Other: placebo — 200 mg lozenges containing anhydrous crystalline maltose taken three times per day for 24 weeks
  Other Names: maltose; sugar pill
  Arms: placebo lozenges

SUMMARY:
This is a study to test lozenges of interferon-alpha that are dissolved in the mouth as a treatment of oral warts in HIV-positive adults.

The hypothesis of this study is that interferon-alpha will be safe and that a higher percentage of subjects given interferon-alpha will experience a complete or nearly complete remission of their oral warts compared to subjects given placebo.

DETAILED DESCRIPTION:
Human papilloma virus (HPV) can cause warts to form in the mouth of infected patients, particularly those with reduced immunity such as people infected with HIV. This is a randomized, double-blind, placebo-controlled trial to determine whether interferon-alpha, delivered in low doses via orally dissolving lozenges, can reduce or eliminate these warts in HIV+ subjects who are receiving combination anti-retroviral therapy (HAART). All potential subjects will have their warts examined and measured at a screening visit. A small amount of one wart (i.e. a biopsy) will be removed for microscopic evaluation to confirm HPV infection and a small amount of blood will be collected for testing. Subjects that qualify for entry will return for a baseline visit at which they will be randomized to active or placebo treatment for 24 weeks. Three out of four subjects will receive active treatment in this study. Subjects must return to the clinic every 6 weeks during treatment to have their warts re-examined. At these follow-up visits, subjects will be asked to complete a brief questionnaire regarding any perceived changes in their warts and their overall mouth condition. A small amount of blood will be taken at the final study visit at week 24 to assess the safety of the interferon lozenges.

ELIGIBILITY:
Inclusion Criteria:

* Must have tested positive for HIV.
* Must have two or more warts inside the mouth.
* Must be receiving a standard course of anti-retroviral therapy (HAART).

Exclusion Criteria:

* Must not be receiving oral or injected steroids.
* Must not be taking other drugs for treatment of oral warts.
* Must not have other active HIV-related opportunistic infections.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 59 (Actual)
Dates: Start 2007-02; Primary Completion 2009-09 (Actual); Study Completion 2009-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Deborah Greenspan, BDS, DSc, Principal Investigator — University of California, San Francisco
Locations (12):
- United States (12):
  - University of California, School of Dentistry, San Francisco, California
  - Nova Southeastern University College of Dental Medicine, Fort Lauderdale, Florida
  - Medical College of Georgia School of Dentistry, Augusta, Georgia
  - University of Illinois at Chicago, College of Dentistry, Chicago, Illinois
  - University of Kentucky College of Dentistry, Lexington, Kentucky
  - University of Maryland Baltimore Dental School, Baltimore, Maryland
  - Division of Oral Medicine and Dentistry, Brigham and Women's Hospital, Boston, Massachusetts
  - UMDNJ - New Jersey Dental School, Newark, New Jersey
  - New York University College of Dentistry, New York, New York
  - University of Pennsylvania School of Dental Medicine, Philadelphia, Pennsylvania
  - Baylor College of Dentistry, Dallas, Texas
  - University of Texas Health Science Center at San Antonio, San Antonio, Texas

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Enrollment took place between January 2007 and March 2009 at 10 university-affiliated dental clinics across the US.
Pre-assignment Details: All 59 enrolled subjects were randomized to treatment and took at least 1 dose of assigned study drug.
Period: Overall Study
Arm/Group | IFN Lozenges | Placebo Lozenges
Started | 45 | 14
Completed | 30 | 11
Not Completed | 15 | 3
Not completed — Adverse Event | 1 | 1
Not completed — Lost to Follow-up | 11 | 1
Not completed — Protocol Violation | 1 | 1
Not completed — Withdrawal by Subject | 2 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | IFN Lozenges | Placebo Lozenges | Total
Number analyzed (Participants) | 45 | 14 | 59
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 45 | 14 | 59
  >=65 years | 0 | 0 | 0
Age Continuous [Mean (Standard Deviation); unit: years] | 45.0 (5.05) | 46.6 (5.43) | 45.4 (5.14)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 1 | 6
  Male | 40 | 13 | 53
Region of Enrollment [Number; unit: participants]
  United States | 45 | 14 | 59

OUTCOME MEASURES:

1. Primary Outcome: Change in Total Oral Mucosal Area Covered by Warts.
Description: Number of subjects with a 75% or greater decrease from baseline to week 24 in total oral wart area
Time Frame: 24 weeks, from baseline to the end of treatment
Population: Per protocol
Measure: Number; unit: participants
Arm/Group | IFN Lozenges | Placebo Lozenges
Number analyzed (Participants) | 36 | 12
participants | 11 | 2
Statistical Analysis 1: Comparison: IFN Lozenges vs Placebo Lozenges; Chi-square analysis of the proportion of subjects in each group meeting the definition of positive response; Test type: Superiority or Other; p = 0.30, Chi-squared

2. Secondary Outcome: Total Surface Area of the Lips Covered by Warts
Description: Number of subjects with a 75% or greater decrease from baseline to week 24 in total lip wart area
Time Frame: 24 weeks, from baseline to the end of treatment
Population: Per protocol - only a sub-set of subjects had lip warts at study entry
Measure: Number; unit: participants
Arm/Group | IFN Lozenges | Placebo Lozenges
Number analyzed (Participants) | 13 | 4
participants | 5 | 0
Statistical Analysis 1: Comparison: IFN Lozenges vs Placebo Lozenges; Chi-square analysis of the proportion of subjects in each group meeting the definition of positive response; Test type: Superiority or Other; p = 0.26, Chi-squared

3. Secondary Outcome: Subject Questionnaire Regarding Changes in Warts
Description: Number of subjects reporting change in oral warts from baseline to week 24 as "better." Scale was subjective with 3 choices: "better," "worse," or "unchanged."
Time Frame: 24 weeks, from baseline to the end of treatment
Measure: Number; unit: participants
Arm/Group | IFN Lozenges | Placebo Lozenges
Number analyzed (Participants) | 36 | 12
participants | 18 | 4
Statistical Analysis 1: Comparison: IFN Lozenges vs Placebo Lozenges; Chi-square analysis of the proportion of subjects in each group reporting change in oral warts from baseline to week 24 as "better."; Test type: Superiority or Other; p = 0.50, Chi-squared

4. Secondary Outcome: Subject Questionnaire Regarding Global Oral Changes
Description: Number of subjects reporting change in global oral health from baseline to week 24 as "better." Scale was subjective with 3 choices: "better," "worse," or "unchanged."
Time Frame: 24 weeks, from baseline to end of treatment
Measure: Number; unit: participants
Arm/Group | IFN Lozenges | Placebo Lozenges
Number analyzed (Participants) | 36 | 12
participants | 14 | 2
Statistical Analysis 1: Comparison: IFN Lozenges vs Placebo Lozenges; Chi-square analysis of the proportion of subjects in each group reporting change in global oral health from baseline to week 24 as "better."; Test type: Superiority or Other; p = 0.29, Chi-squared

5. Secondary Outcome: Investigator Assessment Regarding Changes in Warts
Description: Number of subjects with improvement in oral warts from baseline to week 24 as rated by the attending investigator. Scale was subjective with 3 choices: "improved," "worsened," or "unchanged."
Time Frame: 24 weeks, from baseline to the end of treatment
Measure: Number; unit: participants
Arm/Group | IFN Lozenges | Placebo Lozenges
Number analyzed (Participants) | 36 | 12
participants | 13 | 5
Statistical Analysis 1: Comparison: IFN Lozenges vs Placebo Lozenges; Chi-square analysis of the proportion of subjects rated as "improved" with respect to changes in oral warts from baseline to week 24 by the attending investigator; Test type: Superiority or Other; p = 0.74, Chi-squared

6. Secondary Outcome: Investigator Assessment Regarding Global Oral Changes.
Description: Number of subjects with improvement from baseline to week 24 in global oral health as rated by the attending investigator. Scale was subjective with 3 choices: "improved," "worsened," or "unchanged."
Time Frame: 24 weeks, from baseline to the end of treatment
Measure: Number; unit: participants
Arm/Group | IFN Lozenges | Placebo Lozenges
Number analyzed (Participants) | 36 | 12
participants | 9 | 2
Statistical Analysis 1: Comparison: IFN Lozenges vs Placebo Lozenges; Chi-square analysis of the proportion of subjects rated as "improved" with resepect to changes from baseline to week 24 in global oral health by the attending investigator; Test type: Superiority or Other; p = .71, Chi-squared

ADVERSE EVENTS:
Time Frame: 6 months
Arm/Group | IFN Lozenges | Placebo Lozenges
Serious Adverse Events (participants affected / at risk) | 3/45 | 1/14
Other Adverse Events (participants affected / at risk) | 7/45 | 3/14
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | IFN Lozenges (N=45) | Placebo Lozenges (N=14)
pneumonia (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0)
anal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
asthma (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
esophageal ulcer (Gastrointestinal disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | IFN Lozenges (N=45) | Placebo Lozenges (N=14)
diarrhea (Gastrointestinal disorders) | 3 (3) | 0 (0)
tooth extraction (Surgical and medical procedures) | 3 (3) | 0 (0)
candidiasis (Infections and infestations) | 3 (5) | 1 (1)
upper respiratory tract infection (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 2 (2)

LIMITATIONS AND CAVEATS:
Only 59 of 80 planned subjects were randomized, so statistical power of the study was limited.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less